CLINICAL TRIAL: NCT05173532
Title: The Prescriptive Validity of a Novel Fall Risk Clinical Prediction Rule for People With COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Christopher Brown, Principal Investigator, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-FY2021-1
Record Dates: First submitted 2021-02-19; First posted 2021-12-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Balance; Falls; Fall Risk; Aerobic Exercise; Strength Training; Fall Prevention; Stretching Exercise; Breathing Exercise; Randomized Controlled Trial; Clinical Prediction Rule; Minimal Clinically Important Difference
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients will be blinded to their group assignment. At the time of their group assignment, they will be told that they are in either group "A" (which is actually the experimental group receiving balance training) or "B" (which is actually the active control group receiving the breathing and stretching exercise program), and that both groups may lead to better balance, neither are expected to worsen balance, and it is uncertain which one is more effective at improving balance. After their study participation, patients will guess which group they were in, then told if they guessed correctly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training (Experimental): Static and dynamic balance and gait stability training exercises are performed with supervision by a physical therapist or physical therapist assistant for 30 minutes, 3 times per week, for 8 weeks.
  Interventions: Other: Balance Training
- Breathing and Stretching Exercises (Active Comparator): Patients perform static stretches for all major muscle groups while performing diaphragmatic breathing with supervision by a physical therapist or physical therapist assistant for 30 minutes, 3 times per week, for 8 weeks.
  Interventions: Other: Breathing and Stretching Exercises

INTERVENTIONS:
Other: Balance Training — static and dynamic balance and gait stability exercises
  Arms: Balance Training
Other: Breathing and Stretching Exercises — static stretching while performing diaphragmatic breathing
  Arms: Breathing and Stretching Exercises

SUMMARY:
This study has 3 objectives: (1) demonstrate the effectiveness of balance training for people with COPD, (2) determine which patients with COPD respond best to balance training, and (3) calculate clinically meaningful changes in balance for patients with COPD.

DETAILED DESCRIPTION:
After receiving a detailed explanation of the study, including its risks and benefits, and providing informed consent, patients will be screened for eligibility criteria during a single 75-minute evaluation for participation in a physical therapy based pulmonary rehabilitation program. Those meeting eligibility criteria will be randomly assigned in blocks of four (by clinical site) in a single-blind manner (patients) in a 1:1 ratio to either balance training or a breathing and stretching exercise program. Both groups will receive respiratory muscle stretch exercises, aerobic exercise, strength training, and fall prevention education. The intervention phase will last 8 weeks, with patients being seen 3 times per week for 75 minute sessions supervised by a physical therapist or physical therapist assistant.

ELIGIBILITY:
Inclusion Criteria:

* having reported a fall in the past 5 years, or a near fall in the past year, or a score ≥ 9 on the Short Version of the Falls Efficacy Scale - International Version
* age ≥ 60 years
* both sexes
* spirometrically-confirmed COPD of all disease severity stages
* being independently ambulatory with or without a gait aid
* medical clearance by a physician to participate in pulmonary rehabilitation
* provision of informed consent.

Exclusion Criteria:

* having suffered a recent, severe COPD exacerbation (recent is 30 days or less prior to the study baseline)
* participation in a formal exercise program in the three months prior to the study baseline
* an inability by the patient to complete all study testing due to physical, psychological, communication-barrier, or other unanticipated reasons.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Balance Evaluation Systems Test total score baseline to 4 weeks | 4 weeks
  8-item balance test battery, each item rated from 0-3 then summed for total score, items #3 and #4 are tested on both the right and left side. (#1) HIP/TRUNK LATERAL STRENGTH, (#2) FUNCTIONAL REACH FORWARD, (#3) SINGLE-LEG STANCE, (#4) COMPENSATORY STEPPING CORRECTION- LATERAL, (#5) STAND ON FOAM, EYES CLOSED: (3) 30s stable (2) 30s unstable (1) < 30s (0) Unable, (#6) TIMED "GET UP & GO"
Change in Brief Balance Evaluation Systems Test total score baseline to 8 weeks | 8 weeks
  8-item balance test battery, each item rated from 0-3, then summed for total score, items #3 and #4 are tested on both the right and left side. (#1) HIP/TRUNK LATERAL STRENGTH, (#2) FUNCTIONAL REACH FORWARD, (#3) SINGLE-LEG STANCE, (#4) COMPENSATORY STEPPING CORRECTION- LATERAL, (#5) STAND ON FOAM, EYES CLOSED: (3) 30s stable (2) 30s unstable (1) < 30s (0) Unable, (#6) TIMED "GET UP & GO"

SECONDARY OUTCOMES:
Global Rating of Change in Balance after 4 weeks | 4 weeks
  11-point self-report outcome rating balance improvement(+) or decline(-). Ratings: (+/-5)="very large", (+/-4)="large", (+/-3)="medium", (+/-2)="small", (+/-1)="very small", (0)="none"
Global Rating of Change in Balance after 8 weeks | 8 weeks
  11-point self-report outcome rating balance improvement(+) or decline(-). Ratings: (+/-5)="very large", (+/-4)="large", (+/-3)="medium", (+/-2)="small", (+/-1)="very small", (0)="none"

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A Brown, PT, DPT, Principal Investigator — Texas Woman's University
Locations (3):
- United States (3):
  - Breathing Center of Houston, Houston, Texas
  - Breathing Center of Houston, Sugar Land, Texas
  - Breathing Center of Houston, Webster, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beauchamp MK, Janaudis-Ferreira T, Parreira V, Romano JM, Woon L, Goldstein RS, Brooks D. A randomized controlled trial of balance training during pulmonary rehabilitation for individuals with COPD. Chest. 2013 Dec;144(6):1803-1810. doi: 10.1378/chest.13-1093. PMID 23975185
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Buist AS, McBurnie MA, Vollmer WM, Gillespie S, Burney P, Mannino DM, Menezes AM, Sullivan SD, Lee TA, Weiss KB, Jensen RL, Marks GB, Gulsvik A, Nizankowska-Mogilnicka E; BOLD Collaborative Research Group. International variation in the prevalence of COPD (the BOLD Study): a population-based prevalence study. Lancet. 2007 Sep 1;370(9589):741-50. doi: 10.1016/S0140-6736(07)61377-4. PMID 17765523
- [Background] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management and Prevention of Chronic Obstructive Lung Disease 2017 Report: GOLD Executive Summary. Respirology. 2017 Apr;22(3):575-601. doi: 10.1111/resp.13012. Epub 2017 Mar 7. PMID 28150362
- [Background] Moon Y, Sosnoff JJ. Safe Landing Strategies During a Fall: Systematic Review and Meta-Analysis. Arch Phys Med Rehabil. 2017 Apr;98(4):783-794. doi: 10.1016/j.apmr.2016.08.460. Epub 2016 Aug 31. PMID 27592402
- [Background] Burton E, Farrier K, Lewin G, Petrich M, Boyle E, Hill KD. Are interventions effective in improving the ability of older adults to rise from the floor independently? A mixed method systematic review. Disabil Rehabil. 2020 Mar;42(6):743-753. doi: 10.1080/09638288.2018.1508509. Epub 2018 Dec 4. PMID 30512983
- [Background] Avin KG, Hanke TA, Kirk-Sanchez N, McDonough CM, Shubert TE, Hardage J, Hartley G; Academy of Geriatric Physical Therapy of the American Physical Therapy Association. Management of falls in community-dwelling older adults: clinical guidance statement from the Academy of Geriatric Physical Therapy of the American Physical Therapy Association. Phys Ther. 2015 Jun;95(6):815-34. doi: 10.2522/ptj.20140415. Epub 2015 Jan 8. PMID 25573760
- [Background] Lahousse L, Verlinden VJ, van der Geest JN, Joos GF, Hofman A, Stricker BH, Brusselle GG, Ikram MA. Gait patterns in COPD: the Rotterdam Study. Eur Respir J. 2015 Jul;46(1):88-95. doi: 10.1183/09031936.00213214. Epub 2015 Feb 19. PMID 25700390
- [Background] Morlino P, Balbi B, Guglielmetti S, Giardini M, Grasso M, Giordano C, Schieppati M, Nardone A. Gait abnormalities of COPD are not directly related to respiratory function. Gait Posture. 2017 Oct;58:352-357. doi: 10.1016/j.gaitpost.2017.08.020. Epub 2017 Aug 18. PMID 28866454
- [Background] Horak FB, Wrisley DM, Frank J. The Balance Evaluation Systems Test (BESTest) to differentiate balance deficits. Phys Ther. 2009 May;89(5):484-98. doi: 10.2522/ptj.20080071. Epub 2009 Mar 27. PMID 19329772
- [Background] Shumway-Cook A, Horak FB. Assessing the influence of sensory interaction of balance. Suggestion from the field. Phys Ther. 1986 Oct;66(10):1548-50. doi: 10.1093/ptj/66.10.1548. No abstract available. PMID 3763708
- [Background] Horak FB, Henry SM, Shumway-Cook A. Postural perturbations: new insights for treatment of balance disorders. Phys Ther. 1997 May;77(5):517-33. doi: 10.1093/ptj/77.5.517. PMID 9149762
- [Background] Horak FB. Postural orientation and equilibrium: what do we need to know about neural control of balance to prevent falls? Age Ageing. 2006 Sep;35 Suppl 2:ii7-ii11. doi: 10.1093/ageing/afl077. PMID 16926210
- [Background] de Vries EA, Caljouw SR, Coppens MJ, Postema K, Verkerke GJ, Lamoth CJ. Differences between young and older adults in the control of weight shifting within the surface of support. PLoS One. 2014 Jun 3;9(6):e98494. doi: 10.1371/journal.pone.0098494. eCollection 2014. PMID 24892646
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Rasool J, George K. The impact of single-leg dynamic balance training on dynamic stability. Phys Ther Sport. 2007;8(4):177-184.
- [Background] Sakamoto K, Endo N, Harada A, Sakada T, Tsushita K, Kita K, Hagino H, Sakai A, Yamamoto N, Okamoto T, Liu M, Kokaze A, Suzuki H. Why not use your own body weight to prevent falls? A randomized, controlled trial of balance therapy to prevent falls and fractures for elderly people who can stand on one leg for </=15 s. J Orthop Sci. 2013 Jan;18(1):110-20. doi: 10.1007/s00776-012-0328-3. Epub 2012 Nov 9. PMID 23138409
- [Background] Maki BE, McIlroy WE. The role of limb movements in maintaining upright stance: the "change-in-support" strategy. Phys Ther. 1997 May;77(5):488-507. doi: 10.1093/ptj/77.5.488. PMID 9149760
- [Background] Okubo Y, Schoene D, Lord SR. Step training improves reaction time, gait and balance and reduces falls in older people: a systematic review and meta-analysis. Br J Sports Med. 2017 Apr;51(7):586-593. doi: 10.1136/bjsports-2015-095452. Epub 2016 Jan 8. PMID 26746905
- [Background] Gerards MHG, McCrum C, Mansfield A, Meijer K. Perturbation-based balance training for falls reduction among older adults: Current evidence and implications for clinical practice. Geriatr Gerontol Int. 2017 Dec;17(12):2294-2303. doi: 10.1111/ggi.13082. Epub 2017 Jun 16. PMID 28621015
- [Background] Mansfield A, Wong JS, Bryce J, Knorr S, Patterson KK. Does perturbation-based balance training prevent falls? Systematic review and meta-analysis of preliminary randomized controlled trials. Phys Ther. 2015 May;95(5):700-9. doi: 10.2522/ptj.20140090. Epub 2014 Dec 18. PMID 25524873
- [Background] McCrum C, Gerards MHG, Karamanidis K, Zijlstra W, Meijer K. A systematic review of gait perturbation paradigms for improving reactive stepping responses and falls risk among healthy older adults. Eur Rev Aging Phys Act. 2017 Mar 2;14:3. doi: 10.1186/s11556-017-0173-7. eCollection 2017. PMID 28270866
- [Background] Abellan van Kan G, Rolland Y, Andrieu S, Bauer J, Beauchet O, Bonnefoy M, Cesari M, Donini LM, Gillette Guyonnet S, Inzitari M, Nourhashemi F, Onder G, Ritz P, Salva A, Visser M, Vellas B. Gait speed at usual pace as a predictor of adverse outcomes in community-dwelling older people an International Academy on Nutrition and Aging (IANA) Task Force. J Nutr Health Aging. 2009 Dec;13(10):881-9. doi: 10.1007/s12603-009-0246-z. PMID 19924348
- [Background] Cahalin LP, Braga M, Matsuo Y, Hernandez ED. Efficacy of diaphragmatic breathing in persons with chronic obstructive pulmonary disease: a review of the literature. J Cardiopulm Rehabil. 2002 Jan-Feb;22(1):7-21. doi: 10.1097/00008483-200201000-00002. PMID 11839992
- [Background] Cramer H, Haller H, Klose P, Ward L, Chung VC, Lauche R. The risks and benefits of yoga for patients with chronic obstructive pulmonary disease: a systematic review and meta-analysis. Clin Rehabil. 2019 Dec;33(12):1847-1862. doi: 10.1177/0269215519860551. Epub 2019 Jul 29. PMID 31353959
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] McCarthy B, Casey D, Devane D, Murphy K, Murphy E, Lacasse Y. Pulmonary rehabilitation for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2015 Feb 23;2015(2):CD003793. doi: 10.1002/14651858.CD003793.pub3. PMID 25705944
- [Background] Beauchamp MK, Harrison SL, Goldstein RS, Brooks D. Interpretability of Change Scores in Measures of Balance in People With COPD. Chest. 2016 Mar;149(3):696-703. doi: 10.1378/chest.15-0717. Epub 2016 Jan 12. PMID 26203790
- [Background] Pedersen AB, Mikkelsen EM, Cronin-Fenton D, Kristensen NR, Pham TM, Pedersen L, Petersen I. Missing data and multiple imputation in clinical epidemiological research. Clin Epidemiol. 2017 Mar 15;9:157-166. doi: 10.2147/CLEP.S129785. eCollection 2017. PMID 28352203
- [Background] Austin PC, Steyerberg EW. Events per variable (EPV) and the relative performance of different strategies for estimating the out-of-sample validity of logistic regression models. Stat Methods Med Res. 2017 Apr;26(2):796-808. doi: 10.1177/0962280214558972. Epub 2014 Nov 19. PMID 25411322
- [Result] Ito M, Kakizaki F, Tsuzura Y, Yamada M. Immediate effect of respiratory muscle stretch gymnastics and diaphragmatic breathing on respiratory pattern. Respiratory Muscle Conditioning Group. Intern Med. 1999 Feb;38(2):126-32. doi: 10.2169/internalmedicine.38.126. PMID 10225667
- [Result] Garvey C, Bayles MP, Hamm LF, Hill K, Holland A, Limberg TM, Spruit MA. Pulmonary Rehabilitation Exercise Prescription in Chronic Obstructive Pulmonary Disease: Review of Selected Guidelines: AN OFFICIAL STATEMENT FROM THE AMERICAN ASSOCIATION OF CARDIOVASCULAR AND PULMONARY REHABILITATION. J Cardiopulm Rehabil Prev. 2016 Mar-Apr;36(2):75-83. doi: 10.1097/HCR.0000000000000171. PMID 26906147